CLINICAL TRIAL: NCT02659397
Title: A Study to Assess the Pharmacokinetics, Pharmacodynamics and Safety of Adding ETC-1002 180 mg to Atorvastatin 80 mg Background Therapy in Statin-Treated Patients
Brief Title: A Study Of Pharmacokinetics, Pharmacodynamics And Safety Of Adding ETC-1002 To Atorvastatin 80 mg
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1002-035
Record Dates: First submitted 2016-01-12; First posted 2016-01-20 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Hyperlipidemia
Keywords: LDL-cholesterol; Hypercholesterolemia; ETC-1002; Adenosine triphosphate citrate lyase; Atorvastatin
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ETC-1002 + Atorvastatin (Experimental): ETC-1002 180 mg treatment, oral once daily added-on to Atorvastatin 80 mg once daily
  Interventions: Drug: ETC-1002; Drug: Atorvastatin
- Placebo + Atorvastatin (Placebo Comparator): Placebo treatment, oral once daily added-on to Atorvastatin 80 mg once daily
  Interventions: Drug: Atorvastatin; Drug: Placebo

INTERVENTIONS:
Drug: ETC-1002 — Blinded ETC-1002 180 mg tablet once daily for 4 weeks (Weeks 1 to 4)
  Other Names: bempedoic acid
  Arms: ETC-1002 + Atorvastatin
Drug: Atorvastatin — Atorvastatin 80 mg tablet once daily for 8 weeks (Weeks -4 to 4)
Drug: Placebo — Blinded ETC-1002-matched placebo tablet once daily for 4 weeks (Weeks 1 to 4)
  Arms: Placebo + Atorvastatin

SUMMARY:
The purpose of this research study is to measure the amount of atorvastatin and ETC-1002 in the blood, to determine how ETC-1002 affects the level of LDL-cholesterol (bad cholesterol) and other markers of health and disease in blood and urine, and to see how ETC-1002 is tolerated in the body compared to placebo when added to stable atorvastatin 80 mg background therapy in statin-treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Taking daily stable statin doses for at least 4 weeks prior to screening visit.
* LDL-C between 100-220 mg/dL for patients taking daily high-intensity statin (for 4 weeks prior to switching to sponsor -provided atorvastatin 80 mg/day and stopping all other lipid-regulating drugs and supplements) at the screening visit; or,
* LDL-C between 115-220 mg/dL for patients taking moderate- or low-intensity statin (for 4 weeks prior to switching to sponsor -provided atorvastatin 80 mg/day and stopping all other lipid-regulating drugs and supplements) at the screening visit.
* Must be willing to discontinue other lipid-regulating therapies during the study

Exclusion Criteria:

* History of acute significant cardiovascular disease.
* Current clinically significant cardiovascular disease.
* History of inability to tolerate any statin at any dose due to muscle-related pain or weakness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) pharmacokinetics of atorvastatin and its active metabolites | 2 weeks
  Fold change in Cmax from prior-to to following 2 week treatment with ETC-1002
24-hour area under the curve (AUC) pharmacokinetics of atorvastatin and its active metabolites | 2 weeks
  Fold change in AUC from prior-to to following 2 week treatment with ETC-1002
Percent change in LDL-cholesterol | 4 weeks
  Percent Change from baseline to 4 week treatment, incremental lowering of LDL-C

SECONDARY OUTCOMES:
Percent change in hsCRP | 4 weeks
  Percent change from baseline to following 4 week treatment with ETC-1002
Percent change in total cholesterol | 4 weeks
  Percent change from baseline to following 4 week treatment with ETC-1002
Percent change in non-HDL-cholesterol | 4 weeks
  Percent change from baseline to following 4 week treatment with ETC-1002
Percent change in apolipoprotein B | 4 weeks
  Percent change from baseline to following 4 week treatment with ETC-1002
24-hour post dose plasma concentration pharmacokinetics of ETC-1002 and its active metabolite | 2 weeks
  Fold change in trough exposure from prior-to to following 2 week treatment with ETC-1002

CONTACTS AND LOCATIONS:
Overall Officials: Mary McGowan, MD, Study Director — Esperion Therapeutics, Inc.
Locations (19):
- United States (19):
  - Anaheim, California
  - Los Angeles, California
  - Northridge, California
  - Clearwater, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Port Orange, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Springfield, Illinois
  - Louisville, Kentucky
  - Berlin, New Jersey
  - Rapid City, South Dakota
  - Carrollton, Texas
  - West Jordan, Utah
  - Arlington, Virginia
  - Lynchburg, Virginia
  - Richmond, Virginia
  - Renton, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thompson PD, Rubino J, Janik MJ, MacDougall DE, McBride SJ, Margulies JR, Newton RS. Use of ETC-1002 to treat hypercholesterolemia in patients with statin intolerance. J Clin Lipidol. 2015 May-Jun;9(3):295-304. doi: 10.1016/j.jacl.2015.03.003. Epub 2015 Mar 19. PMID 26073387
- [Background] Nikolic D, Mikhailidis DP, Davidson MH, Rizzo M, Banach M. ETC-1002: a future option for lipid disorders? Atherosclerosis. 2014 Dec;237(2):705-10. doi: 10.1016/j.atherosclerosis.2014.10.099. Epub 2014 Oct 31. PMID 25463109
- [Background] Filippov S, Pinkosky SL, Newton RS. LDL-cholesterol reduction in patients with hypercholesterolemia by modulation of adenosine triphosphate-citrate lyase and adenosine monophosphate-activated protein kinase. Curr Opin Lipidol. 2014 Aug;25(4):309-15. doi: 10.1097/MOL.0000000000000091. PMID 24978142
- [Background] Gutierrez MJ, Rosenberg NL, Macdougall DE, Hanselman JC, Margulies JR, Strange P, Milad MA, McBride SJ, Newton RS. Efficacy and safety of ETC-1002, a novel investigational low-density lipoprotein-cholesterol-lowering therapy for the treatment of patients with hypercholesterolemia and type 2 diabetes mellitus. Arterioscler Thromb Vasc Biol. 2014 Mar;34(3):676-83. doi: 10.1161/ATVBAHA.113.302677. Epub 2014 Jan 2. PMID 24385236
- [Background] Ballantyne CM, Davidson MH, Macdougall DE, Bays HE, Dicarlo LA, Rosenberg NL, Margulies J, Newton RS. Efficacy and safety of a novel dual modulator of adenosine triphosphate-citrate lyase and adenosine monophosphate-activated protein kinase in patients with hypercholesterolemia: results of a multicenter, randomized, double-blind, placebo-controlled, parallel-group trial. J Am Coll Cardiol. 2013 Sep 24;62(13):1154-62. doi: 10.1016/j.jacc.2013.05.050. Epub 2013 Jun 13. PMID 23770179